CLINICAL TRIAL: NCT03940924
Title: Effect of High-Intensity Interval Training Combined With Resistance Training on Body Composition and Gut Microbiota in Postmenopausal Women
Brief Title: HIIT + RT on Body Composition and Gut Microbiota in Postmenopausal Women (PACWOMan)
Acronym: PACWOMan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoire des Adaptations Métaboliques à l'Exercice en conditions Physiologiques et Pathologiques (Other)
Collaborators: CREPS Auvergne Rhône-Alpes (AURA) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018-A03230-55
Record Dates: First submitted 2019-05-02; First posted 2019-05-07 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Overweight; Postmenopausal Women
Keywords: Interval Training; Resistance Training; Overweight; Postmenopausal women; Body composition; Gut microbiota
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant
Masking Description: Data collected on the volunteers will be made anonymous.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Interval Training (HIIT) + Resistance Training (Experimental): Subjects perform three sessions of training during 12 weeks. Session are composed of 20min HIIT program : 60 cycles of speeding up for 8s and pedaling slowly for 12s. (Intensity between 85 and 90% HRmax) + a single set circuits including 10 exercises with a load of 8-12 repetition at around 80% of maximal repetition (1RM)
  Interventions: Other: Training program
- Control Group (No Intervention): Subjects don't have training program. They keep their life style.

INTERVENTIONS:
Other: Training program — High Intensity Interval Training + Resistance Training (HIIT + RT)
  Arms: High Intensity Interval Training (HIIT) + Resistance Training

SUMMARY:
Postmenopausal women, as men, are more prone to central or android obesity than premenopausal women. Recently, some studies have shown that obesity is associated with gut microbiota dysbiosis and gut microbiota could be responsible of fat mass accumulation. Moreover, abdominal fat mass accumulation is associated with an increase of cardiovascular disease risks.

Recent studies suggest that physical activity may positively alter gut microbiota composition. Accumulating evidence suggests that high intensity interval training (HIIT) is an effective strategy for reducing body fat of overweight individuals, especially at the abdominal level. Resistance Training (RT) is associated with increased muscle mass and strength gain in main muscle groups. Thus, RT is also an interesting modality to fight against deconditioning and autonomy loss with age.

The aim of the study was to observed the effects of a 12-week high intensity interval training (HIIT) combined with resistance training (RT) program on gut microbiota and body composition changes in postmenopausal women.

It is hypothesized that HIIT +RT will improve gut microbiota and body composition (including whole body and (intra)-abdominal fat mass) in a concomitant and parallel way.

DETAILED DESCRIPTION:
The aim of the study was to observed the effects of a 12-week high intensity interval training (HIIT) combined with resistance training (RT) program on gut microbiota and body composition changes in postmenopausal women.

30 postmenopausal women will be randomly assigned to HIIT + RT (n= 15) group or Control group (n=15).

HIIT+RT: Each subject performed HIIT protocol consisted of repeated 60 cycles of speeding up for 8 s followed by pedalling slowly for 12 s (20min) Then they performed a single set of 10 exercises with 1 or 2min resting period between exercises. The set consisted of 8-12 repetitions at about 80% maximum repetition (1RM).

Control group : (no training program) Subjects will keep their life style.

Faecal microbiota and body composition will be measured before and after the intervention (3 months).

The investigators will examine the effects of HIIT + RT programs on:

Body composition : total-abdominal and visceral fat mass, total fat free mass and muscle mass Faecal concentration of short chain fatty acids Total fat free mass (and appendicular fat free mass) (DEXA) Glycemic profile (plasma HbA1c, plasma glucose, plasma insulin) Lipid profile (TG, HDL, LDL, total cholesterol) Aerobic capacity (VO2 max) Muscular capacity (fatigability, isometric and dynamic strenght)

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* BMI ≥ 25 and < 40
* Able to follow an exercise protocol
* Eating behavior and physical activity stable since at least 3 month

Exclusion Criteria:

* Subject not able to perform exercise after medical examination
* Subject not able to perform bicycle exercise (pains)
* Use of β-blocker
* Medical treatment that could interfere with the different outcome measures (antibiotics)
* Hormonal Replacement Therapy (HRT)

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Changes in the composition of gut microbiota | Baseline T0 and 3 months after intervention starting
  Evolution of microbiota composition will be evaluated from fecal microbiota analyse before and after intervention.

SECONDARY OUTCOMES:
Total fat mass | Baseline T0 and 3 months after intervention starting
  Change from baseline in total fat mass (g) (estimated from DEXA)
Total fat free mass | Baseline T0 and 3 months after intervention starting
  Change from baseline in total fat free mass (g) (estimated from DEXA)
Abdominal fat mass | Baseline T0 and 3 months after intervention starting
  Change from baseline in abdominal fat mass (g) (estimated from DEXA)
Visceral fat mass | Baseline T0 and 3 months after intervention starting
  Change from baseline in visceral fat mass (g) (estimated from DEXA)
Concentration of Short Chain Fatty Acids (SCFAs) | Baseline T0 and 3 months after intervention starting
  Short Chain Fatty Acid's concentration in faeces will be measured
Evolution of fasting glucose level | Baseline T0 and 3 months after intervention starting
  Change from baseline in plasma fasting glucose level
Evolution of insulinemia | Baseline T0 and 3 months after intervention starting
  Change from baseline in plasma fasting insulinemia (mmol/L)
Evolution of HbA1c | Baseline T0 and 3 months after intervention starting
  Change from baseline in plasma HbA1c (%)
Evolution of lipid profile | Baseline T0 and 3 months after intervention starting
  Change from baseline in plasma triglycerides, total cholesterol, LDL- and HDL cholesterol.
Evolution of plasma inflammatory marker | Baseline T0 and 3 months after intervention starting
  Change from baseline in plasma C-Reactive Protein
Evolution of fitness level | Baseline T0 and 3 months after intervention starting
  Change from baseline in VO2max
Evolution of muscular capacity | Baseline T0 and 3 months after intervention starting
  Change from baseline maximal isometric strenght
Evolution of muscular capacity | Baseline T0 and 3 months after intervention starting
  Change from baseline maximal dynamic strenght

CONTACTS AND LOCATIONS:
Overall Officials: Claire MOREL, Dr, Principal Investigator — CREPS Auvergne Rhône-Alpes / Vichy
Locations (1):
- CREPS Auvergne Rhône-Alpes / Vichy, Bellerive-sur-Allier, Allier, France

REFERENCES:
- [Derived] Dupuit M, Rance M, Morel C, Bouillon P, Boscaro A, Martin V, Vazeille E, Barnich N, Chassaing B, Boisseau N. Effect of Concurrent Training on Body Composition and Gut Microbiota in Postmenopausal Women with Overweight or Obesity. Med Sci Sports Exerc. 2022 Mar 1;54(3):517-529. doi: 10.1249/MSS.0000000000002809. PMID 34628447